CLINICAL TRIAL: NCT03019484
Title: A Complex Intervention to Promote Breastfeeding Self-efficacy
Brief Title: Synergy, Self-efficacy, Breastfeeding and Care (SInergia, Autoeficacia, Lactancia y Cuidados)
Acronym: SIALAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Complejo Hospitalario de Navarra (Other); Universidad Pública de Navarra (Other)
Responsible Party: Principal Investigator, Olga López-Dicastillo, PhD, University of Navarra
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: NUR-SIALAC
Record Dates: First submitted 2016-12-26; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Breast Feeding; Self Efficacy
Keywords: Self-efficacy; Self Efficacy; Nurses's Role; Professional Role; Clinical Trial; Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention consisted on breastfeeding support at three stages: a) week 28-39 pregnancy: women were provided with written information and watch a breastfeeding self-efficacy enhancing video; b) during hospitalization after birth: based on their responses to the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) questionnaire and the observation of a whole breastfeed, nurses provided specific advice using active listening. All the relevant information was registered; c) within one week after birth: a nurse or midwife made a phone call to follow-up mothers breastfeeding behaviour, addressing issues that during the hospitalization needed reinforcement, solving any question or matter that they had and providing positive reinforcement.
  Interventions: Behavioral: Breastfeeding support
- Control: Standard Care (No Intervention): This group received standard antenatal and postnatal care by midwives and nurses caring for them during their regular antenatal visits and after delivery.
  The professionals delivering the intervention were the same than those providing the standard care. That was the reason to first collect the data from the control group and after that organising the training of health professionals to deliver de intervention.

INTERVENTIONS:
Behavioral: Breastfeeding support — Self-efficacy
  Other Names: SIALAC
  Arms: Intervention

SUMMARY:
The aim of the study was to evaluate the effectiveness of a breastfeeding self-efficacy promotion intervention. More specifically our objectives were to: explore changes in self-efficacy following the intervention; explore changes in the initiation and maintenance of breastfeeding following the intervention.

DETAILED DESCRIPTION:
Breastfeeding is the optimal choice for feeding infants in order to ensure a healthy growth and development. Although breastfeeding has many benefits for the infant and the mother, breastfeeding rates drop drastically during the first three months after birth. There is a number of factors that influence the initiation and maintenance of breastfeeding. One of the key factors is maternal self-efficacy in relation to breastfeeding. The aim of the study was the development and evaluation of an intervention to enhance maternal perceived self-efficacy in order to contribute positively to the initiation and maintenance of breastfeeding. This was done by using a complex intervention approach (MRC framework) to design and assess a multi-center controlled trial, involving midwives and nurses working at the Complejo Hospitalario de Navarra (CHN) of the Servicio Navarro de Salud and at the Clínica Universidad de Navarra (CUN). These health professionals were trained to deliver the intervention. The intervention was focused on self-efficacy related aspects and took place at three instances with every mother: in the final stage of pregnancy, during the maternal hospital stay after giving birth, and in the first days after discharge. The participants in the control group received the standard care as provided in each health institution.

ELIGIBILITY:
Inclusion Criteria:

* Intention to breastfeed and no contraindication to do so
* Speak Spanish
* Give informed consent

Exclusion Criteria:

* Unwillingness to breastfeed
* Preterm birth (at <37 weeks gestation)
* Breastfeeding contraindication (galactosemia)
* Breastfeeding-related especial situations (multiple birth; newborn weight <2000g; leporine lip; newborn in intensive care unit)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Changes on Breastfeeding status reported by mothers | at 4 time points: after birth while in hospital (T1); and 4 weeks (T2); 8 weeks (T3); and 6 months (T4) after birth
  The mothers reported whether they were breastfeeding or not.
Changes on maternal breastfeeding self-efficacy measured using the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) questionnaire | at 4 time points: after birth while in hospital (T1); and 4 weeks (T2); 8 weeks (T3); and 6 months (T4) after birth
  The mothers completed the questionnaire in person in T1 and by phone in T2, T3 and T4

CONTACTS AND LOCATIONS:
Overall Officials: Elena Antoñanzas, MSc,BSc,RN, Principal Investigator — Complejo Hospitalario de Navarra; Olga Lopez-Dicastilo, PhD,MSc,BSc, Principal Investigator — University of Navarra
Locations (4):
- Spain (4):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Departamento de Ciencias de la Salud. Universidad Pública de Navarra, Pamplona, Navarre
  - Facultad de Enfermería. Universidad de Navarra, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: No